CLINICAL TRIAL: NCT00950443
Title: Acoustic Reflection Method and Work of Breathing : Two New Methods to Measure Children's Upper Airway Obstruction
Brief Title: Acoustic Reflection Method and Work of Breathing
Acronym: MAVAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P 080606
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-08

CONDITIONS: Airway Obstruction
Keywords: Upper airway obstruction; child; acoustic reflection method; endoscopy; work of breathing; sleep study; CT scan
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Children with upper airway obstruction
  Interventions: Device: Acoustic method and breathing/endoscopic evaluation
- 2 (Active Comparator): Children without upper airway obstruction
  Interventions: Device: Acoustic reflection method

INTERVENTIONS:
Device: Acoustic reflection method — Acoustic reflection gives the longitudinal cross-sectional area profile along airway.Based on planar acoustic wave propagating in a rigid duct connected to airway.
  Arms: 2
Device: Acoustic method and breathing/endoscopic evaluation — Endoscopic evaluation done under general anaesthesia.
  Arms: 1

SUMMARY:
Upper airway obstruction (UAO) is very common in children. Presently, the importance of the UAO is evaluated by the physician during an endoscopic evaluation under general anaesthesia.

The aim of the study is to evaluate two new techniques to quantify the importance of the UAO in children; the acoustic reflection method and the measurement of the work of breathing.

80 children will be included in this monocentric, prospective, open labelled study.

DETAILED DESCRIPTION:
The following evaluations will be performed the day prior to the endoscopic evaluation :1) calculation of a clinical score based on the diurnal and nocturnal respiratory and nutritional tolerance of the UAO, 2) evaluation of the importance and the localisation of the UAO assessed by the acoustic reflection method, 3) measurement of the work of breathing, 4) recording of nocturnal gas exchange during at least 6 hours by s single monitor (Sentec™) which measures pulse oximetry (SaO2) and transcutaneous carbon dioxide (PtcCO2), and evaluation of sleep quality by actigraphy (recording of patient's movements by an Actiwatch™).

All the patients will be re-assessed after 3 months. If no treatment is required, a second clinical evaluation with an acoustic reflection examination will be performed. If a surgical treatment or a noninvasive positive pressure ventilation will be necessary, a second complete evaluation will be performed with an endoscopic examination, the calculation of the clinical score, an acoustic reflection examination, the measurement of the work of breathing, and the recording of the nocturnal gas exchange and sleep quality. This second endoscopic examination will be performed only for medical purpose and not for research only.

The study will last 24 months, comprising 21 months for the inclusion of the patients and 3 months for the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* children aged 0 to 15 years old,
* in a stable state,
* presenting an UAO which requires an endoscopic evaluation under general anaesthesia
* signed informed consent
* affiliation to french health benefits

Exclusion Criteria:

* UAO due solely to a hypertrophy of the adenoids and/or the tonsils,
* patients with a tracheostomy or a non operated cleft palate

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To compare the importance and the localisation of the UAO assessed by the acoustic reflection method and by the endoscopic evaluation under general anaesthesia | At the inclusion visit

SECONDARY OUTCOMES:
To evaluate the feasibility of the acoustic method for the evaluation of UAO in children | At the inclusion visit
To compare the importance and the localisation of the UAO assessed by the acoustic reflection method with the respiratory (during sleep and wakefulness) and nutritional consequences of the UAO | At the inclusion visit
To compare the importance of the UAO assessed by the acoustic reflection method with the measurements of the work of breathing | At the inclusion visit
To compare the importance and the localisation of the UAO assessed by the acoustic reflection method with the results of a high resolution computed tomography scan of the upper airways if done for the medical reasons | At the inclusion visit
To correlate the importance and the localisation of the UAO assessed by the acoustic reflection method with the outcome of surgery if required | At the inclusion and 3 months visits

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas LEBOULANGER, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hospital Armand Trousseau, Pediatric Pulmonology department and ENT department, Paris, France